CLINICAL TRIAL: NCT01287559
Title: Monitoring Necrotizing Enterocolitis in Premature Infants Using Depth-Resolved Broad Spectrum NIRS
Brief Title: Monitoring Necrotizing Enterocolitis in Premature Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Spectros Corporation (Industry)
Collaborators: University of California (Other); University of Texas (Other)
Responsible Party: David Benaron, MD, Spectros Corporation
Other Study IDs: NEO-005
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: NEC; Premature Infant
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with NEC: Infants in which a possible diagnosis of NEC is suspected
- Control Infants: Age-matched and illness-severity matched to NEC subjects, controls are infants NOT suspected of having NEC.

SUMMARY:
The investigators are studying a disease called "necrotizing enterocolitis" (or "NEC" for short), which affects premature infants. It is the most common surgical emergency involving neonates admitted to Newborn Intensive Care Units. Currently, clinicians are unable to identify which infants will go on to develop NEC before they become ill. Clinical signs of illness occur relatively late in the course of the condition, making NEC more difficult to treat. The investigators will test a new probe that uses safe levels of visible and infrared light, with and without ultrasound imaging, to see if the investigators can identify infants before they get sick using a simple, noninvasive test, This test will be repeated through at least one feeding (which stresses the gut) each day. If successful, the health benefit will be large, as it is estimated that treating NEC alone (not including treating its later complications) adds $650 million to the annual health bill.

DETAILED DESCRIPTION:
In this 5-year study, we extend our prior feasibility study to test the hypothesis that very-low-birth-weight neonates (VLBW) who develop necrotizing enterocolitis (NEC) can be reliably detected early in the process using broadband optical spectroscopy sensitive to changes in perfusion of the gut. Such perfusion changes result in regional tissue hypoxemia, which we have demonstrated to be detectable by combined broadband visible/near-infrared tissue oximetry, a real-time method that can assess the adequacy of deep tissue oxygenation. Initially this will be an optical-only device; then combining it with ultrasound will be studied in years 2-5, first on the benchtop, and then in the intensive care unit.

Necrotizing enterocolitis (NEC) is the most common life-threatening surgical emergency encountered in the neonatal intensive care unit [ ]. NEC is a multi-factorial (infectious, inflammatory, and ischemic) disease of the gastrointestinal (GI) tract of newborns and neonates. The end result is mucosal injury and/or transmural necrosis of the intestine. Currently, there is no test to diagnose NEC in the early stages of the disease, before the later and ominous clinical signs appear. The mortality of NEC ranges from 10% to 50%, approaching 100% for neonates with severe forms of the disease characterized by full-thickness necrosis of the intestine, followed by rupture and sepsis.

Ninety percent of NEC cases occur in infants born before 36 weeks' gestational age, occurring in up to 10% of all very-low-birth-weight (VLBW, <1500g) neonates [ ]. A diagnosis of NEC increases the NICU length of stay by 22-60 days, and increases the total hospital charges by $76,000-$186,000 per case [ ]. Finally, Neonates recovering from NEC often incur additional serious complications (malnutrition, liver dysfunction). NEC requiring surgery carries increased risk of cerebral palsy, cognitive or psychomotor impairment, or both.

Repeated attempts to use clinical signs to reliably identify neonates most likely to progress to severe NEC have been unsuccessful. Broadband oximetry appears to offer a solution. Developed by the PI and others, broadband oximetry is sensitive to ischemia. It differs from typical near-infrared spectroscopy (NIRS) methods that generally use only 2-4 wavelengths in that broadband oximetry measures hundreds of wavelengths. Broadband approaches, have shown significantly tighter normal ranges, lower noise, and better reproducibility in vivo. Further, typical NIRS fails to account for shifts in water, fat, blood volume, and stool, any of which can affect oxygenation measurements if not specifically accounted for, making NIRS unreliable for quantitative studies of the gut. In contrast, in our just-completed 1-year feasibility R43 trial, we demonstrated that NEC can be detected using broadband methods. The question remains: how will this new device perform clinically in a multicenter study? By incorporating broadband oximetry monitoring into the management of VLBW neonates, we may detect NEC at its earliest stages and prevent the cascade that leads to bowel necrosis. Success should lead quickly to clinical use, as this team has previously developed, received FDA approval for, and commercialized two biomedical devices.

ELIGIBILITY:
Inclusion Criteria:

* Neonates weighing 500-1,500 g on admission
* Neonates eligible for full care and resuscitation as necessary (no parental request for D.N.R.)
* Enrollment within 12h of suspected NEC; scanning within 24h of diagnosis (unless matched control)
* Informed consent

Exclusion Criteria:

* Refusal or withdrawal of consent
* Skin or mucosal integrity disorders, beyond prematurity (e.g. epidermolysis bullosa, herpes simplex)
* Major congenital malformations and gastrointestinal tract malformation precluding initiations of feeds(e.g., congenital obstruction of GI tract, gastroschisis, omphalocele)
* critically ill neonates, who are unlikely to survive

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants hospitalized for prematurity in a Neonatal ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of NEC by Optical vs. Standard Clinical | 2 weeks
  Diagnosis of NEC by Optical vs. Standard Clinical will be compared, to see if optical facilitates an early diagnosis

SECONDARY OUTCOMES:
Time frame of ischemia associated with NEC: Early vs Late | 2 weeks
  Ischemia may be an early or late feature of NEC. If early, it can serve for early diagnosis. If late, it will help with late diagnosis, but not be useful early in the course of disease. There is no clear evidence as to which of these is true.

CONTACTS AND LOCATIONS:
Overall Officials: David Benaron, MD, Principal Investigator — Spectros Corporation
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of Texas, Dallas, Texas